CLINICAL TRIAL: NCT00772759
Title: A Phase I, Randomised, Double-Blind, Placebo-Controlled, Parallel-Group, Single-Centre Study to Investigate the Safety, Tolerability and Pharmacokinetics of Single and Multiple Ascending Doses of AZD3199 Given Once Daily as Inhaled Formulation Via Turbuhaler to Japanese Healthy Men
Brief Title: Assess Safety, Tolerability and PK of AZD3199 in Japanese
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Lars Grundemar, MD, Medical Science Director, AstraZeneca R&D Lund Sweden
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D0570C00005; 2008-004448-35
Record Dates: First submitted 2008-10-14; First posted 2008-10-15 (Estimated); Last update posted 2009-05-05 (Estimated); Status verified 2009-05

CONDITIONS: Healthy
Keywords: AZD3199; Japanese Healthy Volunteers; Phase I study; Single and Multiple Ascending Dose; safety; tolerability; PK

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Dry powder for oral inhalation
  Interventions: Drug: AZD3199 Turbuhaler®
- 2 (Placebo Comparator): Dry powder for oral inhalation
  Interventions: Drug: Placebo Turbuhaler®

INTERVENTIONS:
Drug: AZD3199 Turbuhaler® — 240, 720 and 2160 μ g, single and multiple (o.d. for 12 days)
  Arms: 1
Drug: Placebo Turbuhaler® — single and multiple (o.d. for 12 days)
  Arms: 2

SUMMARY:
The primary objective of the study is to investigate the safety and tolerability of single and multiple once daily ascending doses of AZD3199 delivered as dry powder via the Turbuhaler inhaler in healthy male Japanese subjects by assessment of incidence and nature of adverse events (AEs), clinically significant abnormalities in ECG parameters, blood pressure (BP), pulse rate, lung function parameters, body temperature and laboratory variables (clinical chemistry, haematology and urinalysis). The secondary objectives of the study are to investigate the pharmacokinetics (PK) of single and multiple ascending doses of AZD3199 by assessment of the degree of accumulation, dose proportionality and time linearity in healthy Japanese subjects, and to investigate systemic β 2- adrenoreceptor mediated effects of single and multiple ascending doses of AZD3199 by assessment of potassium and lactate concentrations, tremor and palpitations, heart rate, QTc, pulse rate, blood pressure and FEV1.

ELIGIBILITY:
Inclusion Criteria:

* Be healthy Japanese volunteers, both of the volunteer's parents, and all grandparents must be Japanese. The volunteer must have been born in Japan, have a valid Japanese passport and must not have lived outside Japan for for more than 5 years.
* BMI 18 - 27, Weight 50 - 85 kg
* Be non-smoker or ex-smoker who has stopped smoking (or using other nicotine products) for >6 months prior to study start.
* Clinical normal physical findings

Exclusion Criteria:

* Any clinically significant disease or disorder
* Any clinically relevant abnormal findings in physical examination, clinical chemistry, haematology, urinalysis, vital signs, ECG or lung function at baseline
* Any clinically important abnormalities in rhythm, conduction or morphology of resting ECG that may interfere with the interpretation of QTc interval changes.
* Use of any medication (including OTC), herbal preparations, vitamins or nutritional supplements within 2 weeks prior to Visit 2, except for occasional intake of paracetamol (maximum daily dose of 4 g)

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2008-10; Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Safety/Tolerability - adverse events (AEs), clinically significant abnormalities in ECG parameters, blood pressure (BP), pulse rate, lung function parameters, body temperature and laboratory variables (clinical chemistry, haematology and urinalysis) | During the study

SECONDARY OUTCOMES:
Pharmacokinetic Parameters derived from plasma concentration and optionally urinary excretion of AZD3199. | During residential period
Pharmacodynamic Potassium and lactate concentrations, tremor and palpitations, heart rate, QTc, pulse rate, blood pressure, and forced expiratory volume in one second (FEV1). | During residential period

CONTACTS AND LOCATIONS:
Overall Officials: Ronnie Beboso, Principal Investigator — Chiltern Clinical Research Unit (CCRU).
Locations (1):
- Research Site, Slough, Berkshire, United Kingdom